CLINICAL TRIAL: NCT07036458
Title: An Open-label, Single-dose, Single-period Study Designed to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of 14C Epaminurad in Healthy Male Subjects
Brief Title: To Evaluate the Mass Balance Recovery, Metabolite Profile and Metabolite Identification in Healthy Male Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: JW24104
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-07

CONDITIONS: Healthy Male Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects will receive a single administration of 14C Epaminurad Oral Solution (Other)
  Interventions: Drug: 14C Epaminurad Oral Solution

INTERVENTIONS:
Drug: 14C Epaminurad Oral Solution — Subjects will receive a single administration of 14C Epaminurad Oral Solution

SUMMARY:
To Evaluate the Mass Balance Recovery, Metabolite Profile and Metabolite Identification in Healthy Male Subjects

DETAILED DESCRIPTION:
The following blood, urine and faecal samples will be collected, and assessments performed, at specified time points

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers

Exclusion Criteria:

1. Subjects does not meet the Inclusion Criteria

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-01-09 (Estimated)

PRIMARY OUTCOMES:
Mass balance recovery of total radioactivity in all excreta (urine and faeces) | Baseline to Day 8
  Collection of plasma, urine and faeces samples during time frame point
Metabolite profling and structural identification | Baseline to Day 8
  Collection of plasma, urine and faeces samples during time frame point

CONTACTS AND LOCATIONS:
Overall Officials: McKenzie Litza, Principal Investigator, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Science, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No